CLINICAL TRIAL: NCT03250988
Title: Prevalence of Comorbid Spasticity and Urinary Incontinence in Residents of a Long-Term Care Facility
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, David Charles, Professor and Vice-Chairman of Neurology, Vanderbilt University Medical Center
Other Study IDs: 170963
Record Dates: First submitted 2017-08-08; First posted 2017-08-16 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Spasticity, Muscle; Muscular Diseases; Musculoskeletal Disease; Muscle Hypertonia; Muscle Spasticity; Neuromuscular Manifestations; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations
MeSH Terms: conditions — Muscle Spasticity; Muscular Diseases; Musculoskeletal Diseases; Muscle Hypertonia; Neuromuscular Manifestations; Signs and Symptoms; Nervous System Diseases; Neurologic Manifestations | interventions — Neurologic Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neurological Examination — The subject will undergo elements of the neurological examination during which the movement disorders neurologist will look specifically for the presence of spasticity. If spasticity is found to be present during the examination, the neurologist will rate the severity of the spasticity in all affected limbs and record whether they would recommend treatment for spasticity, and if so, which treatment(s) they believe would be beneficial for the subject.

SUMMARY:
The purpose of this study is to improve spasticity diagnosis through exploration of potential new diagnostic markers for spasticity that can assist in diagnosis and referral.

DETAILED DESCRIPTION:
The aim of this study is to improve spasticity (a form of muscle rigidity) diagnosis through exploration of potential new diagnostic markers for spasticity that can assist in diagnosis and referral. This will be done by assessing the relatedness of comorbid conditions in patients with spasticity. Emphasis will be placed on urinary incontinence, as previous work has suggested a link between the two conditions. An additional aim of this study is to assess health-related quality of life measures in this population. A medical record review will be performed for all consenting participants residing in Tennessee State Veterans' Homes, which is a long-term care facility in Murfreesboro, TN. Participants will also be asked to complete a brief questionnaire assessing their perceived health-related quality of life, physical wellbeing, and mental wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race, aged 18 and above
* Resident of the selected long-term care facility
* The subject, or if appropriate their medical decision maker, is willing and able to provide written informed consent.

Exclusion Criteria:

* Subjects for whom participation in the study may cause medical harm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of comorbid spasticity and urinary incontinence in a long-term care facility | Up to three months after consent is obtained
  Prevalence of spasticity will be determined by recording the presence/absence of spasticity based on the neurological examination performed on all consenting residents of the long-term care facility. Prevalence of urinary incontinence will be determined by medical record review of all consenting residents of the long-term care facility. The research coordinator will report prevalence of comorbid spasticity and incontinence as a descriptive statistic.

SECONDARY OUTCOMES:
Quality of life in residents of a long-term care facility | Up to three months after consent is obtained
  Subjects (if able) will be asked to complete the EQ-5D-5L questionnaire assessing their perceived health-related quality of life. If the subject is unable to complete the EQ-5D-5L questionnaire, the legal medical decision maker or a relative or friend will be asked to complete the EQ-5D-5L proxy to patient questionnaire, assessing the proxy's view of how the subject perceives their health-related quality of life.
Physical and mental well-being in residents of a long-term care facility | Up to three months after consent is obtained
  Subjects (if able) will be asked to complete the EQ-5D-5L questionnaire assessing their physical and mental well-being. If the subject is unable to complete the EQ-5D-5L questionnaire, the legal medical decision maker or a relative or friend will be asked to complete the EQ-5D-5L proxy to patient questionnaire, assessing the proxy's view of how the subject perceives their physical and mental well-being.
Perceived disability in residents of a long-term care facility | Up to three months after consent is obtained
  Subjects (if able) will be asked to complete the EQ-5D-5L questionnaire assessing their perceived disability. If the subject is unable to complete the EQ-5D-5L questionnaire, the legal medical decision maker or a relative or friend will be asked to complete the EQ-5D-5L proxy to patient questionnaire, assessing the proxy's view of how the subject perceives their disability.

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Tennessee State Veterans' Homes, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gracies JM. Pathophysiology of spastic paresis. II: Emergence of muscle overactivity. Muscle Nerve. 2005 May;31(5):552-71. doi: 10.1002/mus.20285. PMID 15714511
- [Background] Thompson AJ, Jarrett L, Lockley L, Marsden J, Stevenson VL. Clinical management of spasticity. J Neurol Neurosurg Psychiatry. 2005 Apr;76(4):459-63. doi: 10.1136/jnnp.2004.035972. No abstract available. PMID 15774425
- [Background] Pfister AA, Roberts AG, Taylor HM, Noel-Spaudling S, Damian MM, Charles PD. Spasticity in adults living in a developmental center. Arch Phys Med Rehabil. 2003 Dec;84(12):1808-12. doi: 10.1016/s0003-9993(03)00368-x. PMID 14669188
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Welmer AK, von Arbin M, Widen Holmqvist L, Sommerfeld DK. Spasticity and its association with functioning and health-related quality of life 18 months after stroke. Cerebrovasc Dis. 2006;21(4):247-53. doi: 10.1159/000091222. Epub 2006 Jan 27. PMID 16446538
- [Background] Bushman W, Steers WD, Meythaler JM. Voiding dysfunction in patients with spastic paraplegia: urodynamic evaluation and response to continuous intrathecal baclofen. Neurourol Urodyn. 1993;12(2):163-70. doi: 10.1002/nau.1930120210. PMID 7920673
- [Background] Marciniak C, O'Shea SA, Lee J, Jesselson M, Dudas-Sheehan D, Beltran E, Gaebler-Spira D. Urinary incontinence in adults with cerebral palsy: prevalence, type, and effects on participation. PM R. 2014 Feb;6(2):110-20; quiz 120. doi: 10.1016/j.pmrj.2013.07.012. Epub 2013 Aug 23. PMID 23978464
- [Background] Durrant J, Snape J. Urinary incontinence in nursing homes for older people. Age Ageing. 2003 Jan;32(1):12-8. doi: 10.1093/ageing/32.1.12. PMID 12540342
- [Background] von Gontard A, de Jong TP, Rantell A, Nieuwhof-Leppink A, Badawi JK, Cardozo L. Do we manage incontinence in children and adults with special needs adequately? ICI-RS 2014. Neurourol Urodyn. 2016 Feb;35(2):304-6. doi: 10.1002/nau.22823. PMID 26872572
- [Background] Chua K, Chuo A, Kong KH. Urinary incontinence after traumatic brain injury: incidence, outcomes and correlates. Brain Inj. 2003 Jun;17(6):469-78. doi: 10.1080/02699050210154268. PMID 12745703
- [Background] Offermans MP, Du Moulin MF, Hamers JP, Dassen T, Halfens RJ. Prevalence of urinary incontinence and associated risk factors in nursing home residents: a systematic review. Neurourol Urodyn. 2009;28(4):288-94. doi: 10.1002/nau.20668. PMID 19191259
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Johnson TM, Ouslander JG, Uman GC, Schnelle JF. Urinary incontinence treatment preferences in long-term care. J Am Geriatr Soc. 2001 Jun;49(6):710-8. doi: 10.1046/j.1532-5415.2001.49146.x. PMID 11454108